CLINICAL TRIAL: NCT02902146
Title: Bougie Use in Emergency Airway Management
Acronym: BEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-4146
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bougie (Active Comparator): On the first intubation attempt, this arm will attempt to place a bougie into the trachea, followed by an endotracheal tube.
  Interventions: Device: Bougie
- No bougie (endotracheal tube first) (Active Comparator): On the first intubation attempt, this arm will attempt to place an endotracheal tube into the trachea directly.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Bougie
  Arms: Bougie
Device: Endotracheal tube
  Arms: No bougie (endotracheal tube first)

SUMMARY:
This prospective, open-label trial randomizes adult patients intubated in the ED with a Macintosh blade to use or not use a bougie for the first intubation attempt. The primary outcome is first pass success.

DETAILED DESCRIPTION:
The primary analysis for all outcomes will be for those with a difficult airway characteristic (defined as any of: cervical immobility, obesity, large tongue, short neck, small mandible, facial or neck trauma, airway edema, blood in the airway, or vomit in the airway).

We will also analyze all outcomes for all patients enrolled, regardless of whether they have a difficult airway characteristic.

We plan to enroll 374 patients with a difficult airway characteristic (DAC). The total enrollment for the trial will be higher, depending on the proportion of patients that have a DAC.

Based on observational data, we aim to detect a 9% absolute difference in first pass success (95% with bougie compared to 86% without the bougie), which requires enrollment of 374 patients with a DAC.

To help achieve balanced randomization for patients with a DAC, patients are stratified into two groups: 1) obese or cervical immobilization present and 2) not obese and no cervical immobilization.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be undergoing orotracheal intubation in the ED with a Macintosh blade (using either video or direct laryngoscopy)
2. The patient must be presumed to be 18 years of age or older at the time of enrollment.

Exclusion Criteria:

1. Known anatomic distortion of the upper airway or perilaryngeal structures.
2. Prisoner or under arrest
3. Known or suspected to be pregnant, based on the opinion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096

RESULTS

PARTICIPANT FLOW:
Groups:
- Bougie: On the first intubation attempt, this arm will attempt to place a bougie into the trachea, followed by an endotracheal tube.
  Bougie
- No Bougie (Endotracheal Tube First): On the first intubation attempt, this arm will attempt to place an endotracheal tube into the trachea directly.
  Endotracheal tube
Period: Overall Study
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Started | 381 | 376
Completed | 381 | 376
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bougie | No Bougie (Endotracheal Tube First) | Total
Number analyzed (Participants) | 381 | 376 | 757
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (18) | 46 (18) | 46 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 121 | 230
  Male | 272 | 255 | 527
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Pass Success
Description: First pass success is defined as placement of the endotracheal tube (ETT) into the trachea on the first attempt. An attempt begins when the laryngoscope enters the mouth, and ends if either of the following occur:
  1. the laryngoscope leaves the mouth, regardless of whether an attempt was made to pass the endotracheal tube or bougie.
  2. if the operator cannot intubate the trachea with the first tube device (ETT or bougie), and switches to any other tube device, even if the laryngoscope blade remains in the mouth.
  A patient will be considered to achieve the primary outcome if they are intubated successfully on the first attempt.
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Number analyzed (Participants) | 381 | 376
Participants | 373 | 328

2. Secondary Outcome: First Pass Success Without Hypoxemia
Description: First pass success without hypoxemia. Hypoxemia is defined as a pulse oximetry value (SpO2) less than 90% at any point during intubation, or a drop of more than 10% from baseline if starting below 90%. The outcome of hypoxemia will be recorded beginning when the first attempt begins and ending one minute after inflation of the ETT cuff.
  A patient will be considered to achieve this outcome if 1) they are intubated successfully on the first attempt, and 2) do not experience hypoxemia on the first attempt.
Time Frame: 5 minutes
Population: The patients not included in this number had no oximetry waveform available
Measure: Count of Participants; unit: Participants
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Number analyzed (Participants) | 371 | 366
Participants | 317 | 282

3. Secondary Outcome: Time to Intubation (First Attempt)
Description: Time to intubation will be defined as the time elapsed between the beginning of the intubation attempt to inflation of the ETT cuff when the tube is in the trachea.
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Number analyzed (Participants) | 381 | 376
seconds | 38 [29 to 51] | 36 [25 to 54]

4. Secondary Outcome: Esophageal Intubation
Description: defined as passage of the ETT into the esophagus, with subsequent ventilation, and then removal. Clinically, esophageal intubation is identified by the absence of end-tidal carbon dioxide, abnormal physical exam, and hypoxia. This does not count passage of the ETT into the esophagus during the attempt if the ETT is removed during the attempt.
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Number analyzed (Participants) | 381 | 376
Participants | 0 | 3

5. Secondary Outcome: Hypoxemia
Description: Hypoxemia is defined as a pulse oximetry value (SpO2) less than 90% at any point during intubation, or a drop of more than 10% from baseline if starting below 90%. The outcome of hypoxemia will be recorded beginning when the first attempt begins and ending one minute after inflation of the ETT cuff.
Time Frame: 5 minutes
Population: The patients not included in these numbers did not have a valid oximetry waveform during intubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
Number analyzed (Participants) | 371 | 364
Participants | 47 | 50

ADVERSE EVENTS:
Time Frame: 5 minutes following intubation
Description: We did not monitor all-cause mortality during the hospital stay, as this trial examined ED intubation.
Arm/Group | Bougie | No Bougie (Endotracheal Tube First)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 12/381 | 11/376
Other Adverse Events (participants affected / at risk) | 47/371 | 50/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bougie (N=381) | No Bougie (Endotracheal Tube First) (N=376)
Cardiac arrest in the ED at any time (Cardiac disorders) | 12 | 11 — All were unrelated to study participation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bougie (N=371) | No Bougie (Endotracheal Tube First) (N=374)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 47 | 50 — Oxygen saturation less than 90 % during or within 1 minute of intubation completion. This outcome only includes participants on whom we were able to record an oxygen saturation during intubation. Therefore, it is less than the total.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02902146/Prot_SAP_000.pdf